CLINICAL TRIAL: NCT04439604
Title: Impact of Body Mass Index on Positive End-Expiratory Pressure Guided by Electrical Impedance Tomography for Patients Under General Anesthesia: A Retrospective Observational Study
Brief Title: Impact of Body Mass Index on Positive End-expiratory Pressure Guided by Electrical Impedance Tomography for Patients Under General Anaesthesia
Acronym: PEPTI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: NOWOBILSKI 2019
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: General Anesthetic; Positive Expiratory Pressure; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient undergoing surgery under general anaesthesia
  Interventions: Other: regional ventilation monitoring

INTERVENTIONS:
Other: regional ventilation monitoring — regional ventilation monitoring

SUMMARY:
The induction of general anaesthesia is associated with a fall in lung volume due in particular to a decrease in muscle tone and the formation of denitrogenation atelectasis. Many recent studies insist on the need to apply a so-called "protective" strategy of intraoperative ventilation, which combines the use of recruitment manoeuvres, reduced tidal volume (Vt) (6-8ml/kg) and positive expiratory pressure (PEEP) to prevent these phenomena. However, the setting of PEEP remains debated and several authors agree on the need to individualize ventilatory parameters, particularly in obese patients, without describing the individualization tools.

In the ICU, it has been shown that electrical impedance tomography (EIT) can be used to individualise the PEEP level in a simple and non-invasive way. Therefore, we wish to determine whether the use of this technique during general anaesthesia allows for the individualization of PEEP, and whether the value determined is correlated with the body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient who received general anesthesia with orotracheal intubation.
* Patient who has undergone surgery of the following types: : abdominal surgery by laparotomy or laparoscopy, emergency or scheduled

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical Patients
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2018-10-06 (Actual); Primary Completion 2019-07-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
electrical impedance tomography | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France